CLINICAL TRIAL: NCT04689178
Title: Cervical Cancer Screening Uptake: A Randomised Controlled Trial Assessing the Effect of Sending Invitation Letters to Nonadherent Women Combined With Sending Their General Practitioners a List of Their Nonadherent Patients
Brief Title: Cervical Cancer Screening Uptake: A Randomised Controlled Trial Assessing the Effect of Sending Invitation Letters to Nonadherent Women
Acronym: IMPACTGP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RC20_0364
Record Dates: First submitted 2020-11-27; First posted 2020-12-30 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer screening; General Practitioner; Organized screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Invitation letter + GP reminder (Arm 1) (Experimental)
  Interventions: Other: Invitation letter + GP reminder
- Invitation letter (Arm 2) (Active Comparator)
  Interventions: Other: Invitation letter
- Usual care (Arm 3) (No Intervention)

INTERVENTIONS:
Other: Invitation letter + GP reminder — 40-65 year-old women who did not perform a PAP test over the last 3 years will receive an invitation to consult a health professional to perform a screening test, AND GPs will receive the list of their 40-65 year-old patients who did not perform a PAP test over the last 3 years
  Arms: Invitation letter + GP reminder (Arm 1)
Other: Invitation letter — 40-65 year-old women who did not perform a PAP test over the last 3 years will receive an invitation to consult a health professional to perform a screening test. GPs will NOT receive any list of their non-adherent patients.
  Arms: Invitation letter (Arm 2)

SUMMARY:
Context:

In France, cervical cancer (CC) screening was opportunistic until recently. The target population includes women aged 25 to 65 years. About 66% of women aged 25-40 years have performed a screening test over the last three years but this figure decreases to 55% in women over 40. The third "Cancer Plan" proposed by the French National Institute for Cancer recommends to achieve an 80% participation in eligible women.

Improving women compliance to CC screening is a major challenge to decrease cancer incidence and mortality.

To improve patient adherence, a CC screening organization will be launched in 2020 at a national scale in France. Women who did not perform a PAP test over the last 3 years will receive an invitation letter from the local public health association in charge of cancer screening organization. The invitation letter will remind women that they should consult a healthcare professional (a general practitioner (GP), a gynecologist or a midwife) to perform a screening test.

Providing GPs with a list of their non-adherent patients could also improve women compliance to CC screening recommendations.

The study objective is to assess whether sending both an invitation letter to non-adherent women and a list of their non-adherent patients to GPs ("invitation letter + GP reminder" group) could increase the proportion of women who perform a screening test, compared to only sending an invitation letter to non-adherent women ("invitation letter" group) or not sending any invitation ("usual care" group).

DETAILED DESCRIPTION:
Design, Setting and Participants:

The investigators will conduct a 3-arm, cluster-randomized, controlled trial in the Loire-Atlantique region, in France.

The study will include a total of 1,500 GPs and about 100,000 women. The randomization will be based on GP practices to avoid a contamination bias resulting from shared tracking mechanisms and communication between GPs within a given practice. Thus, several GPs working in the same practice will be assigned to the same study arm. Women on the patient list of a given GP will be assigned to the arm of this GP.

Intervention:

After a cluster randomization according to the practice, the GPs and their female patients will be included in one of the following 3 arms:

* "Invitation letter + GP reminder" (Arm 1): 40-65 year-old women who did not perform a PAP test over the last 3 years will receive an invitation to consult a health professional to perform a screening test, AND GPs will receive the list of their 40-65 year-old patients who did not perform a PAP test over the last 3 years;
* "Invitation letter" (Arm 2): 40-65 year-old women who did not perform a PAP test over the last 3 years will receive an invitation to consult a health professional to perform a screening test. GPs will NOT receive any list of their non-adherent patients.
* "Usual care" (arm 3): 40-65 year-old women who did not perform a PAP test over the last 3 years will NOT receive any invitation to consult a health professional to perform a screening test. GPs will NOT receive any list of their non-adherent patients.

Expected Results

The investigators expect an increase in the proportion of women who perform a screening test in the intervention arm (arm 1), compared to arms 2 and 3. Previous studies have suggested that the proportion of women adherent to CC screening could be increased by 25% in arm 1 compared to arm 3, whereas the participation could be increased by 15% in arm 2 compared to arm 3.

Considering that the proportion of adherent women in arm 3 should be of about 55%, the absolute increase in participation could reach 11% in arm 1, and 6.6% in arm 2.

A higher adherence to CC screening could improve the detection of pathological lesions by 5% for pathological pap smears and by 10% for positive HPV tests.

ELIGIBILITY:
Inclusion Criteria for GPs:

- All GPs practicing in the Loire-Atlantique region (Western France) will be included.

Inclusion criteria for patients :

* women aged 40 to 65 years,
* being on the patient list of the GPs participating in the study,
* living in the Loire-Atlantique region (Western France),
* being affiliated to the National Health Insurance.

Exclusion Criteria for GPs:

- GPs who could refuse to participate by contacting the research team.

Inclusion criteria for patients :

* Refusal to participate to the study
* Female patients who underwent total hysterectomy and those who received a pathological result of a previous pap smear (asc-us or CIN) are not eligible to participate in the CC screening and therefore excluded from the study.
* Women not registered with a GP located in Loire-Atlantique will not be included.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195000 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of women aged 40-65 who performed a screening test (HPV test or PAP smear) over the last 3 years, 6 months after the intervention | 6 months

SECONDARY OUTCOMES:
Description of the types of screening tests carried out in first intention | 6 months
  Proportion of cytological tests performed among all screening tests
Description of the types of screening tests carried out in first intention | 6 months
  Proportion of HPV tests performed among all screening tests
Description of the results of screening tests carried out in first intention | 6 months
  Proportion of abnormal test results (cytology, HPV) among all screening tests performed
Description of the types of tests performed for follow-up of lesions detected | 6 months
  Proportion of "reflex" tests performed (number of cervical smears after a positive HPV result) among abnormal test results
Description of the types of tests performed to follow lesions detected by screening | 12 months
  Proportion of biopsies and conizations performed among abnormal screening test results
Description the results of the tests performed to follow lesions detected by screening | 12 months
  Proportion of high-grade lesions detected (second, a third-grade cervical intraepithelial neoplasia, including in situ carcinomas and cancers) among the abnormal screening tests
Description of the treatments undergone by the women following abnormal screening tests | 12 months
  Percentages of treatments performed (conization, laser, hysterectomy) among the abnormal screening tests
Description of the factors associated with lower participation in screening | 6 months
  Participation rate according to age (over 50), income (women with low incomes qualifying for basic health coverage) and comorbidities.
Description of the healthcare trajectory of women undergoing a screening test | 6 months
  Proportion of women who resort to a GP, a midwife or a gynaecologist to undergo their screening test

CONTACTS AND LOCATIONS:
Overall Officials: Cedric RAT, Professor, Principal Investigator — Nantes University Hospital; Anne-Sophie BANASZUK, Doctor, Principal Investigator — Centre de coordination des dépistages des cancers (CRCDC)
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teigne D, Banaszuk AS, Grimault C, Abes L, Gaultier A, Rat C. Cervical cancer screening uptake: A randomized controlled trial assessing the effect of sending invitation letters to non-adherent women combined with sending their general practitioners a list of their non-adherent patients (study protocol). Front Public Health. 2022 Nov 10;10:1035288. doi: 10.3389/fpubh.2022.1035288. eCollection 2022. PMID 36438208